CLINICAL TRIAL: NCT03259750
Title: Validity and Reliability of the Foot and Ankle Ability Measure Turkish Version for Athletes
Brief Title: The Foot and Ankle Ability Measure (FAAM) is Translated From English to Turkish and Assess the Validity and Reliability in Athletic Population Who Have Foot and Ankle Disorders.
Status: Completed | Type: Observational
Sponsor: Serkan Usgu (Other)
Responsible Party: Sponsor-Investigator, Serkan Usgu, Assistant Professor of Physiotherapy and Rehabilitation, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Other Study IDs: HEK09/103
Record Dates: First submitted 2017-08-14; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Ankle; Injury, Superficial, Multiple (With Foot)
Keywords: Self-reported outcome instrument; Sport; Ankle and foot; Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- professional athletes: athlete who volunteered in this study that should be a member of a professional sport team, All athletes must complete self reported outcome instrument (FAAM-T)
  Interventions: Other: Foot and Ankle Ability Measure Turkish version (FAAM-T) questionnaire

INTERVENTIONS:
Other: Foot and Ankle Ability Measure Turkish version (FAAM-T) questionnaire — Self reported outcome instrument

SUMMARY:
Sport activity induces a relevant risk for lower extremities especially ankle and foot structures. Athletes who participate in basketball, volleyball and soccer are predisposed. Self-reported outcome instruments have been used by clinicians to assess the treatment interventions effectiveness directed at patients with pathologies and identify impairments, disabilities and quality of life. The assessment of musculoskeletal injuries can be problem without clinical, radiological examination and on scores from patient-based questionnaires. The information from these questionnaires provides us good evidence if there is not interpretation of obtained scores. The Foot and Ankle Ability Measure (FAAM) is a self-reported outcome instrument for patients with foot and ankle disorders available in English, German, and French. The FAAM has a sports subscale and activity of daily living (ADL) subscale that can assess the activities that requires higher level. The aim of this study is to translate the FAAM into Turkish language, perform a cross-cultural adaptation, and investigate the reliability, validity of the translated version in athletic population

ELIGIBILITY:
Inclusion Criteria:

1. Participants should be professional athletes
2. Age ranges must be 18-40 years old
3. Clinical diagnosis of ankle and foot injury

   1. Acute condition
   2. Chronic condition
4. Injuries must to happened in sport activities.

Exclusion Criteria:

1. If athletes had injuries to hip, knee, lower leg within the previous 6 months before the study.
2. The history of surgery to the above-mentioned areas.
3. Coexisting musculoskeletal injuries in other body parts, or chronic conditions.

   1. Systematic diseases
   2. Neurological or vascular conditions.
   3. Alcohol abuse
   4. Psychiatric disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The professional Turkish-speaking athletes who foot and ankle disorders participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2009-08-20 (Actual); Primary Completion 2014-05-20 (Actual); Study Completion 2015-07-12 (Actual)

PRIMARY OUTCOMES:
FAAM-T questionnaire | 3 days
  The FAAM-T is comprised of separately scored 21-item Activity of Daily Living (ADL) and 8-item Sports subscales. Each item is scored on a five-point Likert scale from 4 to 0, item score totals can be varied from 0 to 84 for the ADL and from 0 to 32 for the sports subscale. The percentage scores calculated with the total score of each subscale is divided by the highest potential score and multiplied by 100.

SECONDARY OUTCOMES:
Visual Analogue Scale | 3 days
  Visual analogue scale (VAS) is used to represent pain and also functional limitation in sport. The VAS includes numbers, words, figures, to recognize the patients rate the pain or functional limitation level. Responses were converted to numerical scores by measuring the distance from the zero point to the vertical mark. This distance was recorded to the nearest millimeter.
6 meters shuttle run | 3 days
  Participants sprinted up and back twice along a 6 meters course. Participants were required to start with one leg forward on the start line. Time started from the initial forward movement of the athlete and stopped when the athlete crossed the line. Each participants was timed with a hand-held stopwatch and recorded in second.
Triple forward hop | 3 days
  Participants were asked to face parallel down the test "runway," and, when signaled, participant hopped as far as possible in the forward direction with 3 consecutive hops on the same leg. The distance between the starting line and the place where participant lands on the third hop measured at the heel was recorded in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Usgu, PhD, Principal Investigator — Hasan Kalyoncu University; Yavuz Yakut, Prof, Study Chair — Hasan Kalyoncu University; Sıdıka Fatma Uygur, Prof, Study Director — Cyprus International University; Gunseli Usgu, PhD, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 6 months after publication

REFERENCES:
- [Background] Gonzalez-Sanchez M, Li GZ, Ruiz Munoz M, Cuesta-Vargas AI. Foot and ankle ability measure to measure functional limitations in patients with foot and ankle disorders: a Chinese cross-cultural adaptation and validation. Disabil Rehabil. 2017 Oct;39(21):2182-2189. doi: 10.1080/09638288.2016.1219772. Epub 2016 Sep 6. PMID 27597231
- [Result] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Result] Carcia CR, Martin RL, Drouin JM. Validity of the Foot and Ankle Ability Measure in athletes with chronic ankle instability. J Athl Train. 2008 Apr-Jun;43(2):179-83. doi: 10.4085/1062-6050-43.2.179. PMID 18345343
- [Result] Borloz S, Crevoisier X, Deriaz O, Ballabeni P, Martin RL, Luthi F. Evidence for validity and reliability of a French version of the FAAM. BMC Musculoskelet Disord. 2011 Feb 8;12:40. doi: 10.1186/1471-2474-12-40. PMID 21303520
- [Result] Moreira TS, Magalhaes Lde C, Silva RD, Martin RL, Resende MA. Translation, cross-cultural adaptation and validity of the Brazilian version of the Foot and Ankle Ability Measure questionnaire. Disabil Rehabil. 2016 Dec;38(25):2479-90. doi: 10.3109/09638288.2015.1137979. Epub 2016 Feb 15. PMID 26878102
- [Result] Hoch JM, Legner JL, Lorete C, Hoch MC. The Validity of the Quick-FAAM in Patients Seeking Treatment for an Acute or Subacute Foot or Ankle Health Condition. J Sport Rehabil. 2017 May 1;26(3):jsr.2016-0089. doi: 10.1123/jsr.2016-0089. Epub 2016 Sep 16. PMID 27633016
- [Result] Arunakul M, Arunakul P, Suesiritumrong C, Angthong C, Chernchujit B. Validity and Reliability of Thai Version of the Foot and Ankle Ability Measure (FAAM) Subjective Form. J Med Assoc Thai. 2015 Jun;98(6):561-7. PMID 26219160
- [Result] Weel H, Zwiers R, Azim D, Sierevelt IN, Haverkamp D, van Dijk CN, Kerkhoffs GM. Validity and reliability of a Dutch version of the Foot and Ankle Ability Measure. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1348-54. doi: 10.1007/s00167-014-3480-9. Epub 2014 Dec 25. PMID 25536950
- [Result] Uematsu D, Suzuki H, Sasaki S, Nagano Y, Shinozuka N, Sunagawa N, Fukubayashi T. Evidence of validity for the Japanese version of the foot and ankle ability measure. J Athl Train. 2015 Jan;50(1):65-70. doi: 10.4085/1062-6050-49.3.42. Epub 2014 Oct 13. PMID 25310247
- [Result] Sartorio F, Vercelli S, Bravini E, Bargeri S, Moroso M, Plebani G, Ferriero G. [Foot and ankle ability measure: cross-cultural translation and validation of the Italian version of the ADL module (FAAM-I/ADL)]. Med Lav. 2014 Jul 15;105(5):357-65. Italian. PMID 25134631
- [Result] Donahue M, Simon J, Docherty CL. Critical review of self-reported functional ankle instability measures. Foot Ankle Int. 2011 Dec;32(12):1140-6. doi: 10.3113/FAI.2011.1140. PMID 22381198
- [Result] Martin RL, Irrgang JJ. A survey of self-reported outcome instruments for the foot and ankle. J Orthop Sports Phys Ther. 2007 Feb;37(2):72-84. doi: 10.2519/jospt.2007.2403. PMID 17366962
- [Result] Arnold BL, Wright CJ, Ross SE. Functional ankle instability and health-related quality of life. J Athl Train. 2011 Nov-Dec;46(6):634-41. doi: 10.4085/1062-6050-46.6.634. PMID 22488189
- [Result] Hoch JM, Druvenga B, Ferguson BA, Houston MN, Hoch MC. Patient-Reported Outcomes in Male and Female Collegiate Soccer Players During an Athletic Season. J Athl Train. 2015 Sep;50(9):930-6. doi: 10.4085/1062-6050-50.5.03. Epub 2015 Jul 24. PMID 26207439